CLINICAL TRIAL: NCT03500718
Title: Changes in the Threshold of Electrically Evoked Compound Action Potential in Children Following Cochlear Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Principal Investigator, Dr. Aparna Das, JUNIOR RESIDENT, Jawaharlal Institute of Postgraduate Medical Education & Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JIP/IEC/2017/0339
Record Dates: First submitted 2018-04-02; First posted 2018-04-18 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Cochlear Hearing Loss
Keywords: cochlear implant; threshold of electrically evoked compound action potential; neural response telemetry
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric patients with bilateral sensorineural hearing loss (Experimental): One group will be studied: Patients undergoing cochlear implantation surgery between age 1 and 6 years who meet the above inclusion and exclusion criteria seen in JIPMER during the study period.
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant — After cochlear implantation, cochlear nerve is stimulated by giving a current over the electrodes placed in the cochlea and the current is measured by electrically evoked Compound Action Potential (ECAP).

SUMMARY:
After cochlear implantation, cochlear nerve is stimulated by giving a current over the electrodes placed in the cochlea and the current is measured by electrically evoked Compound Action Potential (ECAP).This ECAP is measured intra operatively, after 4 weeks( at switch on), after 3months and 6 months following cochlear implantation.

DETAILED DESCRIPTION:
After cochlear implantation, cochlear nerve is stimulated by giving a current over the electrodes placed in the cochlea and the current is measured by electrically evoked Compound Action Potential (ECAP).This ECAP is measured intra operatively, 4 weeks(at switch on) and after 3months and 6 months following cochlear implantation. Neural Response Telemetry (NRT) is a quick and non-invasive way of recording ECAP of the peripheral auditory nerves in-situ. It gives clinicians valuable information for programming the T- (Threshold) and C-(Comfort) - levels of the recipient's speech processor map. Intraoperative NRT in conjunction with electrode impedance data can help indicate the integrity of the implanted electrodes and the electrode/auditory nerve interface, confirming that the implant is functioning correctly intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* All children between 1 and 6 years of age undergoing cochlear implantation in JIPMER during the study period.

Exclusion Criteria:

* Incomplete electrode array insertion.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in threshold of ECAP after cochlear implantation. | during implantation, at switch on( 4 weeks), after 3months and 6months.
  To evaluate changes in threshold of ECAP during cochlear implantation, at switch on( 4 weeks), after 3 months and 6 months following cochlear implantation.

SECONDARY OUTCOMES:
Correlate the amplitude of ECAP with T & C levels. | 2 years
  Correlating the amplitude of ECAP with threshold and comfortable levels and creating a MAP.
Correlate amplitude of ECAP with cochlear nerve diameter measured pre-operatively. | 2 mins
  By correlating amplitude of ECAP with cochlear nerve diameter we can determine the site to be operated preoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- JIPMER, Puducherry, India

IPD SHARING:
Plan to Share IPD: No
Confidentiality regarding patient's participation in the study will be maintained throughout the study period as well as after completion of the study.

REFERENCES:
- [Background] Kim JR, Abbas PJ, Brown CJ, Etler CP, O'Brien S, Kim LS. The relationship between electrically evoked compound action potential and speech perception: a study in cochlear implant users with short electrode array. Otol Neurotol. 2010 Sep;31(7):1041-8. doi: 10.1097/MAO.0b013e3181ec1d92. PMID 20634770
- [Background] van Eijl RH, Buitenhuis PJ, Stegeman I, Klis SF, Grolman W. Systematic review of compound action potentials as predictors for cochlear implant performance. Laryngoscope. 2017 Feb;127(2):476-487. doi: 10.1002/lary.26154. Epub 2016 Nov 2. PMID 27804133